CLINICAL TRIAL: NCT05231694
Title: Specific Stimulation Mode Electroacupuncture Combined With NGF for Recovery Period of Ischemic Stroke：Protocol for a Randomized Controlled Clinical Trial
Brief Title: The Impact of Electroacupuncture Combined With NGF on Clinical Effect and Functional Changes on Ischemic Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Ningbo No.2 Hospital (Other); second people hospital of lishui (Unknown)
Responsible Party: Principal Investigator, Xianming Lin, Clinical Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XLin
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; Convalescence; Electroacupuncture; nerve growth factor
MeSH Terms: conditions — Ischemic Stroke; Convalescence; Hereditary Sensory and Autonomic Neuropathies | interventions — Nerve Growth Factor; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- sham EA + placebo group (Other): sham EA + placebo group contain sham EA intervention and placebo injection
  Interventions: Drug: Placebo injection; Device: sham EA intervention
- sham EA + NGF group (Other): sham EA + NGF group contain sham EA intervention and NGF injection
  Interventions: Drug: Nerver growth factor (NGF) injection; Device: sham EA intervention
- EA + placebo group (Other): EA + placebo group contain EA intervention and placebo injection
  Interventions: Drug: Placebo injection; Device: EA intervention
- EA + NGF group (Other): EA + NGF group contain EA intervention and NGF injection
  Interventions: Drug: Nerver growth factor (NGF) injection; Device: EA intervention

INTERVENTIONS:
Drug: Nerver growth factor (NGF) injection — The 20ug nerve growth factor (NO.S20060051, Jinlujie) will be obtained from Hiteck Biopharmaceutical Co., Ltd, Wuhan, China. mNGF will be dissolved in 1 ml sterile water for injection and then injected intramuscularly at gluteal muscle, once a day for 4 weeks. Dose modification is not allowed for mNGF.
  Arms: EA + NGF group; sham EA + NGF group
Drug: Placebo injection — The patients will receive 1ml volume of physiological saline (PS) injected into the gluteal muscle, once a day for 4 weeks.
  Arms: EA + placebo group; sham EA + placebo group
Device: EA intervention — Patients take supine position. After skin disinfection with 75% ethanol routine disinfection, the stainless needle (size 0.25mm×40mm, Hua Tuo brand, Suzhou Medical Supplies Company Ltd in Jiangsu, China) will be inserted in GV20（Baihui) and the stainless needle(size 0.25mm×25mm, described above) will be inserted in GV26 (Shuigou), acupoints will be stimulated manually until patients feel soreness, distension or heaviness (the reaction of "De Qi"). Then, the needles are stimulated by using an acupuncture point nerve stimulator (HANS-200, Nanjing Jinsheng, Ltd., China) with a frequency of 2/100 Hz and an intensity of 3 mA for 40 min (a homemade relay cycled power to the electrode for 6 sec on and 6 sec off), 28 days as a course of treatment, once a day.
  Arms: EA + NGF group; EA + placebo group
Device: sham EA intervention — The only difference between sham EA intervention and EA intervention is that the stimulator is connected to the needle handle without power for 40 min intervention.
  Arms: sham EA + NGF group; sham EA + placebo group

SUMMARY:
Ischemic stroke is a common clinical disease, often accompanied by motor dysfunction and cognitive impairment. At present, clinical treatment for patients with ischemic stroke recovery is limited and ineffective. The emergence of NGF has surprised the field of neurorehabilitation, but the clinical effect is not satisfactory. The main problem is that NGF is a macromolecular material with a molecular weight of 13.4 KD, which is difficult to penetrate the blood brain barrier. A large number of previous studies in our team have found that electroacupuncture with specific stimulation mode can open the blood brain barrier and induce NGF into the brain。Therefore, the purpose of this study is to investigate the effect of specific stimulation mode electroacupuncture combined with NGF treatment together with rehabilitation training on patients with ischemic stroke recovery period and to explore the mechanism of this combination therapy to improve brain function, which creates a new method and theoretical basis for nerve rehabilitation of integrated traditional Chinese and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

* people with first-ever ischemic stroke confirmed by CT or/and MRI;
* 14 days to 6 months after stroke onset;
* 50 years≤aged≤80 years;
* 3≤modified Rankin Score (mRS)≤4, and Mini-Mental State Examinations (MMSE)<27;
* Patients can accept treatment with EA and have good compliance;
* Patients have clear consciousness, pain perception and resolution ability to complete basic communication;
* willing to participate and be randomized to one of the groups.

Exclusion Criteria:

* transient ischemic attack, subarachnoid hemorrhage, cerebral hemorrhage and other cerebrovascular diseases;
* severe heart, liver, kidney dysfunction and severe coagulation dysfunction;
* cerebral infarction caused by repeated recurrence of stroke, brain surgery or trauma, and brain tumors;
* severe neurological deficits before stroke, such as visual and auditory impairment, aphasia, agnosia, severe hemiplegia, or affected limb function before stroke, such as cerebral palsy, polio, fracture, and mRs≥1;
* diseases with affecting cognitive function such as congenital dementia, or alcohol, drug or substance abuse;
* lactation, pregnancy or intend to be pregnant within 6 months;
* needlesickness, needle phobia and skin infection at acupuncture site;
* pacemaker, implantable cardioverter defibrillator carriers or conductive metallic foreign bodies in the body;
* allergy to NGF;
* currently enrolled in another clinical trial or participation in other clinical trials within the last 3 months.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
basic cure rate | end of treatment (week 4)
  patients with the modified Rankin Score ≤ 2 are judged as basic cure, and basic cure rate= number of patients with the modified Rankin Score ≤ 2 / group * 100 %. The modified Rankin Score ranges from 0 to 6, and the more severe the neurological deficit, the higher the score. at the end of treatment, the modified Rankin Score is recorded in all four groups.

SECONDARY OUTCOMES:
simplified Fugl-Meyer Assessment of motor function score (FMA) | baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  simplified Fugl-Meyer Assessment of motor function score sums up a total score (maximum 100 points ), including an assessment of the upper extremity (maximum 66 points) and lower extremity (maximum 34 points). Improvement in simplified Fugl-Meyer Assessment of motor function score suggests the recovery of motor function
Modified Barthel Index (MBI) | baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  Modified Barthel Index is one of the measures to evaluate activities of daily living and consisted of 10 items (bathing, personal hygiene, feeding, dressing, toilet use, bladder continence, bowel control, stair climbing, chair/bed transfers and mobility. Besides, wheelchair score only if patient is unable to ambulate and is trained in wheelchair managemen). The maximum total score of Modified Barthel Index is 100, with a higher score meaning less dependent to help.
timed up and go test (TUGT) | baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  timed up and go test is an assessment tool for measuring mobility in stroke patients. In the timed up and go test, each patient is asked to stand up from an armchair at height 45 cm, walk a distance of 3 m, turn, walk back to the chair, and sit back down in chair . With interval of one minute rest, a patient is required to repeat the test three times to take its mean for statistical analysis
Tinetti Performance Oriented Mobility Assessment (POMA) | baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  POMA scale can be used to assess the balance with B-POMA including nine components (sitting balance, arises, attempts to arise, immediate standing balance, standing balance, nudged, eyes closed, turning 360 , and sitting down; maximum 16 points) and to evaluate the gait with G-POMA including seven components (initiation of gait, step length, step symmetry, step continuity, path, trunk, and walking stance; maximum 12 points) . A patient with POMA scored less than 24 points suggets balance dysfunction and scored less than 15 points indicates danger of falling.
Montreal Cognitive Assessment (MoCA) | baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  The Montreal Cognitive Assessment is a 30-point test and focuses on assessing seven cognitive domains including visual-spatial and executive abilities, naming, delayed memory recall, attention, abstraction, language and orientation functions . A patient with MoCA scored less than 26 points suggets cognitive impairment.
Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) | baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  Loewenstein Occupational Therapy Cognitive Assessment is a 91-point test to estimate cognitive functions including orientation (8 points), perception (24 points), visual movement organization (28 points), thought operation (27 points), attention and concentration (4 points). The higher the score of patients indicates the better the cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data and results of this study need to be confirmed by Lin Xianming

REFERENCES:
- [Result] Cao Y, Yu S, Zhang Q, Yu T, Liu Y, Sun Z, Zhao M, Wang W, Zhao JZ; Chinese Stroke Association Stroke Council Guideline. Chinese Stroke Association guidelines for clinical management of cerebrovascular disorders: executive summary and 2019 update of clinical management of intracerebral haemorrhage. Stroke Vasc Neurol. 2020 Dec;5(4):396-402. doi: 10.1136/svn-2020-000433. Epub 2020 Dec 1. PMID 33262243
- [Result] Zhao N, Zhang H, Liu T, Liu J, Xiang Y, Shu G, Li C, Xie J, Chen L. Neuromodulatory Effect of Sensorimotor Network Functional Connectivity of Temporal Three-Needle Therapy for Ischemic Stroke Patients with Motor Dysfunction: Study Protocol for a Randomized, Patient-Assessor Blind, Controlled, Neuroimaging Trial. Evid Based Complement Alternat Med. 2021 Jan 4;2021:8820324. doi: 10.1155/2021/8820324. eCollection 2021. PMID 33488759
- [Result] Byun K, Hyodo K, Suwabe K, Ochi G, Sakairi Y, Kato M, Dan I, Soya H. Positive effect of acute mild exercise on executive function via arousal-related prefrontal activations: an fNIRS study. Neuroimage. 2014 Sep;98:336-45. doi: 10.1016/j.neuroimage.2014.04.067. Epub 2014 May 2. PMID 24799137
- [Result] Cope M, Delpy DT. System for long-term measurement of cerebral blood and tissue oxygenation on newborn infants by near infra-red transillumination. Med Biol Eng Comput. 1988 May;26(3):289-94. doi: 10.1007/BF02447083. No abstract available. PMID 2855531
- [Result] Broderick JP, Adeoye O, Elm J. Evolution of the Modified Rankin Scale and Its Use in Future Stroke Trials. Stroke. 2017 Jul;48(7):2007-2012. doi: 10.1161/STROKEAHA.117.017866. Epub 2017 Jun 16. No abstract available. PMID 28626052
- [Result] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Result] Son H, Park C. Effect of turning direction on Timed Up and Go test results in stroke patients. Eur J Phys Rehabil Med. 2019 Feb;55(1):35-39. doi: 10.23736/S1973-9087.18.05202-4. Epub 2018 Jul 6. PMID 29984566
- [Result] Chu JJ, Chen XJ, Shen SS, Zhang XF, Chen LY, Zhang JM, He J, Zhao JF. A poor performance in comprehensive geriatric assessment is associated with increased fall risk in elders with hypertension: a cross-sectional study. J Geriatr Cardiol. 2015 Mar;12(2):113-8. doi: 10.11909/j.issn.1671-5411.2015.02.006. PMID 25870613
- [Result] Zhao W, You H, Jiang S, Zhang H, Yang Y, Zhang M. Effect of Pro-kin visual feedback balance training system on gait stability in patients with cerebral small vessel disease. Medicine (Baltimore). 2019 Feb;98(7):e14503. doi: 10.1097/MD.0000000000014503. PMID 30762779
- [Result] Huang J, Lin Z, Wang Q, Liu F, Liu J, Fang Y, Chen S, Zhou X, Hong W, Wu J, Madrigal-Mora N, Zheng G, Yang S, Tao J, Chen L. The effect of a therapeutic regimen of Traditional Chinese Medicine rehabilitation for post-stroke cognitive impairment: study protocol for a randomized controlled trial. Trials. 2015 Jun 16;16:272. doi: 10.1186/s13063-015-0795-x. PMID 26077459
- [Result] Larsson AC, Palstam A, Persson HC. Physical Function, Cognitive Function, and Daily Activities in Patients Hospitalized Due to COVID-19: A Descriptive Cross-Sectional Study in Sweden. Int J Environ Res Public Health. 2021 Nov 4;18(21):11600. doi: 10.3390/ijerph182111600. PMID 34770113
- [Result] Lu H, Zhang T, Wen M, Sun L. Impact of repetitive transcranial magnetic stimulation on post-stroke dysmnesia and the role of BDNF Val66Met SNP. Med Sci Monit. 2015 Mar 14;21:761-8. doi: 10.12659/MSM.892337. PMID 25770310
- [Result] Cai Y, Zhang CS, Ouyang W, Li J, Nong W, Zhang AL, Xue CC, Wen Z. Electroacupuncture for poststroke spasticity (EAPSS): protocol for a randomised controlled trial. BMJ Open. 2018 Feb 27;8(2):e017912. doi: 10.1136/bmjopen-2017-017912. PMID 29487073
- [Result] Yu KW, Lin CL, Hung CC, Chou EC, Hsieh YL, Li TM, Chou LW. Effects of electroacupuncture on recent stroke inpatients with incomplete bladder emptying: a preliminary study. Clin Interv Aging. 2012;7:469-74. doi: 10.2147/CIA.S37531. Epub 2012 Nov 8. PMID 23152677
- [Result] Baber N. International conference on harmonisation of technical requirements for registration of pharmaceuticals for human use (ICH). Br J Clin Pharmacol. 1994 May;37(5):401-4. doi: 10.1111/j.1365-2125.1994.tb05705.x. No abstract available. PMID 8054244
- [Result] Zhen X, Sun X, Dong H. Health Technology Assessment and Its Use in Drug Policies in China. Value Health Reg Issues. 2018 May;15:138-148. doi: 10.1016/j.vhri.2018.01.010. Epub 2018 May 3. PMID 29729645
- [Derived] Dai M, Zhao Y, Jia Z, Xu S, Xu N, Wu X, Liu J, Wu L, Yu K, Lin X. Effect of Specific mode electroacupuncture stimulation combined with NGF during the ischaemic stroke: Study protocol for a randomized controlled trial. Clinics (Sao Paulo). 2024 Jul 20;79:100451. doi: 10.1016/j.clinsp.2024.100451. eCollection 2024. PMID 39033586